CLINICAL TRIAL: NCT01668121
Title: Pharmacokinetic Study on Budesonide/Formoterol Device-metered Dry Powder Inhalers, Two Batches of Symbicort Turbuhaler and Budesonide/Formoterol Easyhaler: Randomised, Double-blind, Double-dummy, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Study on Budesonide/Formoterol Device-metered Dry Powder Inhalers
Acronym: REFLI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3103012
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort Turbohaler (Experimental): Symbicort Turbohaler
  Interventions: Drug: Symbicort Turbohaler; Drug: Budesonide/formoterol Easyhaler
- Budesonide/formoterol Easyhaler (Active Comparator): Budesonide/formoterol Easyhaler
  Interventions: Drug: Symbicort Turbohaler; Drug: Budesonide/formoterol Easyhaler

INTERVENTIONS:
Drug: Symbicort Turbohaler
Drug: Budesonide/formoterol Easyhaler

SUMMARY:
The primary objective of this study is to evaluate the acceptance range with which two Symbicort Turbohaler batches could be declared bioequivalent in a bioequivalence setting. The secondary objective is to compare pharmacokinetic parameters of the reference product batches and Budesonide/formoterol Easyhaler.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Males and females, 18-55 (inclusive) years of age.
3. Normal weight defined as body mass index (BMI) > 19 and < 30 kg/m2 (BMI= weight/height2).
4. Weight at least 50 kg.
5. Forced expiratory volume in one second (FEV1) at least 80% of the predicted value measured at the screening.
6. Good general health ascertained by detailed medical history, and laboratory and physical examinations.

Exclusion Criteria:

1. Vulnerable subjects (i.e. persons under any administrative or legal supervision).
2. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease within previous 2 years; or evidence of active or quiescent pulmonary tuberculosis, fungal and viral infections in the airways.
3. Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol and ibuprofen for occasional pain are allowed.
4. Intake of any medication that could affect the outcome of the study. As an exception, contraceptives and hormone replacement therapy are allowed. The use of medicines which are strong CYP3A4 inducers or inhibitors are restricted for at least 2 weeks prior to the first study treatment administration and during the study.
5. Any clinically significant abnormal laboratory value or physical finding (including electrocardiogram [ECG] and vital signs) that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study, as judged by the investigator. More specifically, supine HR < 45 or > 100 bpm after 10-min rest or supine systolic BP >140 or < 90 or diastolic BP > 90 or < 60 mmHg after a 10-minute rest, or a QTc-Bazett (QTcB interval) > 450 msec at screening evaluation.
6. Known hypersensitivity to the active substances or the excipient (lactose, which contains small amounts of milk protein) of the drug.
7. History of vasovagal collapses.
8. History of anaphylactic/anaphylactoid reactions.
9. History of seizures including febrile seizures.
10. Pregnant or lactating females.
11. Females of childbearing potential if they are not using proper contraception (mechanical and/or hormonal contraception, intrauterine device [IUD] or surgical sterilization). Double method of contraception is needed when using oral or mechanical contraception: e.g. condom in conjunct with oral contraception and spermicidal product with mechanical contraception (please see section 5.7 for details).
12. Recent or current (suspected) drug abuse or positive result in the drugs abuse test.
13. Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 16 units per week for females [1 unit = 4 cl spirits or equivalent]).
14. Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study (from the screening visit to the end-of-study visit).
15. Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages during the treatment periods until 24 h after study treatment administration.
16. Blood donation or loss of significant amount of blood within 30 days prior to the first study treatment administration.
17. Administration of another investigational drug within 30 days prior to the first study treatment administration.
18. Unsuitable veins for repeated venepuncture or for cannulation.
19. Inability to learn the correct inhalation technique.
20. Predictable poor compliance or inability to communicate well with the study centre personnel.
21. Inability to participate in all treatment periods.
22. The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
23. Positive result in HIV, hepatitis B or C tests.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax of plasma Budesonide concentration | within 12 h
Pharmacokinetic parameter AUCt of plasma Budesonide concentration | within 12 h
Pharmacokinetic parameter Cmax of plasma Formoterol concentration | within 24 h
Pharmacokinetic parameter AUCt of plasma Formoterol concentration | within 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — Parexel; Merja Mäkitalo, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- PAREXEL International GmbH, Berlin, Germany